CLINICAL TRIAL: NCT06973369
Title: The Effect of Education Given With Creative Drama Method Based on Leininger's Theory on the Cultural Sensitivity and Effectiveness Levels of Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Uzeyir SOLAK, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ATASBEUZE001
Record Dates: First submitted 2025-04-17; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Nursing Education; Nursing Students; Creative Drama; Cultural Sensitivity
Keywords: Leininger; Nursing students; Creative drama; Cultural sensitivity; Cultural effectiveness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental)
  Interventions: Other: LEININGER THEORY BASED CREATIVE DRAMA EDUCATION METHOD
- CONTROL (Experimental)
  Interventions: Other: TRADITIONAL EDUCATION METHOD

INTERVENTIONS:
Other: LEININGER THEORY BASED CREATIVE DRAMA EDUCATION METHOD — The effects of Leininger theory-based creative drama training given to nursing students for five weeks on the students' cultural sensitivity and effectiveness levels will be determined.
  Arms: INTERVENTION
Other: TRADITIONAL EDUCATION METHOD — Leininger theory training will be given to nursing students for five weeks and its effects on the students' cultural sensitivity and effectiveness levels will be determined.
  Arms: CONTROL

SUMMARY:
This study aims to determine the effect of cultural care education given with creative drama method according to Leininger theory on the cultural sensitivity and effectiveness levels of nursing students. The study will be conducted as a pre-test and post-test randomized controlled experimental study. The universe of the study consists of fourth-year students (n=80) of "Agri Ibrahim Cecen University, Faculty of Health Sciences, Department of Nursing". In this study, students in the intervention and control groups will be determined by simple randomization method. After the theoretical course content is given based on Leininger theory, students in the intervention group will be given creative drama technique with cases and students in the control group will be given traditional case examples. A pre-test will be applied before the training program and a post-test will be applied after the training program.

ELIGIBILITY:
Inclusion Criteria:

* Want to participate in the study voluntarily,
* Have taken the Intercultural Nursing course,
* Have taken 75% of the practical nursing courses.

Exclusion Criteria:

* Being a nurse working in the clinic,
* Being a foreign national,
* Being in the initiative group and not participating in the creative drama application,
* The student wanting to leave the research at any stage,
* Not filling out the data collection forms or filling them incompletely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cultural Sensitivity Score | At Baseline, Immediately after training
  The participants' level of cultural sensitivity will be assessed using the Cultural Sensitivity Scale. This tool evaluates nursing students' awareness, respect, and responsiveness to cultural diversity in healthcare. The scale will be administered immediately before and after the educational intervention. The difference in scores will indicate the impact of the creative drama-based training grounded in Leininger's Transcultural Nursing Theory.
Change in Intercultural Effectiveness Score | At Baseline, Immediately after training
  The Intercultural Effectiveness Scale will measure the participants' intercultural effectiveness level. This scale assesses communication skills, emotional resilience, and cultural flexibility in cross-cultural interactions. The test will be administered immediately before and after the intervention. The difference in scores will indicate the impact of the creative drama-based training grounded in Leininger's Transcultural Nursing Theory.

CONTACTS AND LOCATIONS:
Locations (1):
- Agri Ibrahim Cecen University, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No